# **Statistical Analysis Plan**

A Phase 1, Randomized, Open-Label, Parallel-Group, Clinical trial protocol title: Relative Bioavailability Study to Investigate the Pharmacokinetics, including Food Effect, as well as the Safety and Tolerability of Single Doses of New Immediate Release Tablet Formulations of Emodepside (BAY 44-4400), compared to Oral Solution, in Healthy Male Subjects HMR code: 17-008 Sponsor code: DNDI-EMO-03 EudraCT no: 2017-003091-31 CRO details: Hammersmith Medicines Research Cumberland Avenue London NW10 7EW Sponsor details: DNDi, Chemin Louis Dunant, 15, 1202 Geneva Switzerland Phone: +41 22 906 9230 Issued: 23 March 2018 Version: 1 Based on: Protocol Version 3, 1 February 2018 Number of pages: 61 Prepared by: Helen Topping

# **Table of contents**

| 1 | LIST | OF ABBREVIATIONS | 5 |
|----|------|-------------------------------------------------------|----|
| 2 | SIGN | NATURES | 7 |
| 3 | INTE | RODUCTION | 8 |
| 4 | STUI | DY OBJECTIVE(S) AND ENDPOINT(S) | 8 |
| | 4.1 | Study Objective(s) | 8 |
| | | 4.1.1 Primary Objective | 8 |
| | | 4.1.2 Secondary Objectives | 8 |
| | 4.2 | Study Endpoint(s) | 9 |
| | | 4.2.1 Primary Endpoint | 9 |
| | | 4.2.2 Secondary Endpoints | |
| | | 4.2.3 Exploratory Endpoints | |
| | 4.3 | Statistical Hypotheses | 9 |
| 5 | STUI | DY DESIGN | 10 |
| 6 | TIM | E AND EVENTS TABLE | 12 |
| 7 | PLA | NNED ANALYSES | 14 |
| | 7.1 | Interim Analyses | 14 |
| | | 7.1.1 Persons responsible for analysis | 14 |
| | 7.2 | Final Analysis | 14 |
| | | 7.2.1 Persons responsible for analysis | |
| 8 | SAM | PLE SIZE CONSIDERATIONS | 15 |
| | 8.1 | Sample Size Assumptions | 15 |
| 9 | ANA | LYSIS POPULATIONS | 15 |
| | 9.1 | Analysis Datasets | 15 |
| 10 | TRE | ATMENT COMPARISONS | 15 |
| 11 | GEN | ERAL CONSIDERATIONS FOR DATA ANALYSES | 16 |
| | 11.1 | Data Display Treatment and Other Subgroup Descriptors | 16 |
| | 11.2 | Conventions for Summary Statistics and Data Displays | 16 |
| 12 | DAT | A HANDLING CONVENTIONS | 17 |
| | 12.1 | Premature Withdrawal and Missing Data | 17 |
| | 12.2 | Derived and Transformed Data | 17 |
| | 12.3 | Assessment Windows | 18 |
| | 12.4 | Values of Potential Clinical Importance | 18 |
| 13 | STUI | DY POPULATION | 18 |
| | 13.1 | Disposition of Subjects | 18 |

| | 13.2 | Protocol Deviations | 19 |
|---|---|---|---|
| | 13.3 | Demographic and Baseline Characteristics | 19 |
| | 13.4 | Treatment Compliance | 19 |
| 14 | SAFI | ETY ANALYSES | 19 |
| | 14.1 | Extent of Exposure | 20 |
| | 14.2 | Adverse Events | 20 |
| | 14.3 | Deaths, Serious Adverse Events and Other Significant Adverse E | events 20 |
| | 14.4 | Adverse Events Leading to Withdrawal from the Study | 21 |
| | 14.5 | Clinical Laboratory Evaluations | 21 |
| | 14.6 | Other Safety Measures | 21 |
| | | 14.6.1 Vital signs | 21 |
| | | 14.6.2 ECG | 21 |
| | | 14.6.3 Physical and neurological examination | 22 |
| 15 | PHA | RMACOKINETIC ANALYSES | 22 |
| | 15.1 | Pharmacokinetic Concentration Data | 22 |
| | 15.2 | Pharmacokinetic Parameters | 23 |
| 16 | REFI | ERENCES | 23 |
| 17 | ATT | ACHMENTS | 24 |
| | 17.1 | Table of Contents for Data Display Specifications | 24 |
| | 17.2 | Data Display Specifications | 29 |
| | | 17.2.1 Table Outlines | 29 |
| | | 17.2.2 Figure Outlines | 40 |
| | | 17.2.3 Listing Outlines | 44 |
| APP | ENDIX | A: LABORATORY RANGES | 55 |
| APP | PENDIX | B: PHARMACOKINETIC ANALYSIS | 57 |
| 1 | CAL | CULATION METHODS | 57 |
| | 1.1 | Data Handling Conventions | 57 |
| | | 1.1.1 Actual vs Planned Times | 57 |
| | | 1.1.2 Missing and BQL Concentrations | 57 |
| | 1.2 | AUC Calculations | 57 |
| | 1.3 | Lambda-z Calculations | 57 |
| | 1.4 | Observed v Predicted Values | 58 |
| 2 | GEN | ERAL CONSIDERATIONS FOR DATA ANALYSIS | 58 |
| | 2.1 | Derived and transformed data | 58 |
| | 2.2 | Summary data | 58 |
| 3 | PAR | AMETER DEFINITIONS | 59 |

| 3.1 | Plasma Parameters | | |
|----------|-------------------|------------------|------|
| | 3.1.1 | Emodepside | . 59 |
| APPENDIX | C: SAI | MPLE PAGE LAYOUT | 61 |

### 1 List of abbreviations

 $\lambda_z$  Terminal rate constant

AE Adverse Event ANOVA Analysis of variance

AUC Area under concentration-time curve

 $AUC_{0-t}$  AUC from time zero to time t

AUC<sub>0-t</sub>/Dose AUC from time zero t to time t, corrected for dose

AUC<sub>0-t,norm</sub> AUC from time zero t to time t, corrected for dose and body weight

AUC<sub>last</sub> AUC from time zero to last measurable concentration

BMI Body Mass Index BP Blood Pressure

BQL Below the limit of quantification

CI Confidence Interval

C<sub>max</sub> Maximum Plasma Concentration

 $C_{max}/Dose$   $C_{max}$  corrected by dose

C<sub>max, norm</sub> C<sub>max</sub> corrected by dose and body weight

CRF Case Report Form CTR Clinical Trial Report ECG Electrocardiogram

HMR Hammersmith Medicines Research

HR Heart Rate

ICH International Conference on Harmonization

IR Immediate Release

LLOQ Lower Limit of Quantification LSF Liquid Service Formulation

MedDRA Medical Dictionary for Regulatory Activities

MRT Mean residence time

MRT<sub>last</sub> Mean residence time at last measurable concentration

N Number of subjects

n Number of observations used in analysis

PCI Potential clinical importance

PK Pharmacokinetic(s)

PR Portion of the ECG from the beginning of the P wave to the beginning of the

QRS complex, representing atrioventricular node function.

Q1 Lower quartile Q3 Upper quartile

QRS The QRS complex of the ECG reflects the rapid depolarization of the right

and left ventricles.

QT Portion of the ECG between the onset of the Q wave and the end of the T

wave, representing the total time for ventricular depolarization and

repolarization.

QTc Corrected portion of the ECG between the onset of the Q wave and the end

of the T wave, representing the total time for ventricular depolarization and

repolarization.

QTcB QTc interval with Bazett's correction method QTcF QTc interval with Fridericia's correction method

RR Portion of the ECG between consecutive R waves, representing the

ventricular rate

| SAP | Statistical Analysis Plan |
|---------------|--------------------------------------|
| SD | Standard deviation |
| SRG | Safety Review Group |
| $t_{1/2}$ | Terminal elimination half-life |
| $t_{1/2,0-t}$ | Dominant half-life |
| TEAE | Treatment-Emergent Adverse Event |
| $t_{max}$ | Time to maximum plasma concentration |

# 2 Signatures

The following persons have read and agreed the content of this Statistical Analysis Plan:

Helen Topping Senior Statistician, HMR

Signature

28 MARZOUS

Dr Jeremy Dennison Principal Investigator, HMR

Signature

28 MAR 2018

Date

Jean-Yves Gillon Head of Translation, DNDi

Signature

27 Rard 2018

Frédéric Monnot Filarial Team Leader, DNDi

Signature

Date

### 3 Introduction

This Statistical Analysis Plan (SAP) is based on the current trial protocol (version 3, 1 February 2018). Where statistical methods differ substantially between this SAP and the protocol, that will be identified in this document.

This SAP describes the datasets and the statistical methods to be used for the reporting and analysis of all data collected during the trial.

The randomisation code will not be broken before this SAP is finalised. If a future protocol amendment necessitates a substantial change to the statistical analysis of the trial data, this SAP will be amended accordingly. If, after database lock, additional analyses are required to supplement the planned analyses described in this SAP, those unplanned analyses will not be described in an amended SAP, but they will be identified in the integrated clinical study report (CSR). Any deviations from this SAP will be documented in the CSR.

This SAP has been written in consideration of the following guidelines:

- International Conference on Harmonization (ICH) E9, Guidance for Industry: Statistical Principles for Clinical Trials (ICH E9 1998)<sup>1</sup>; and
- ICH E3, Guidance for Industry: Structure and Content of Clinical Study Reports (ICH E3 1995)<sup>2</sup>.

Pharmacokinetic analysis will be done using WinNonlin v7 on a Windows PC. Statistical analysis will be done using SAS<sup>®</sup> 9.3 on a Windows PC.

# 4 Study Objective(s) and Endpoint(s)

# 4.1 Study Objective(s)

#### 4.1.1 Primary Objective

To investigate the pharmacokinetics, including relative bioavailability and food effect, of two new immediate release (IR)-tablet formulations of emodepside in comparison to the liquid service formulation (LSF) oral solution.

#### 4.1.2 Secondary Objectives

To investigate and compare safety and tolerability of single oral doses of emodepside formulations in healthy subjects.

### 4.2 Study Endpoint(s)

#### 4.2.1 Primary Endpoint

 Based on the plasma concentration—time data, the following PK parameters of emodepside will be calculated:

o Main: AUC<sub>0-7d</sub>, AUC<sub>0-7d</sub>/Dose, C<sub>max</sub>, C<sub>max</sub>/Dose

#### 4.2.2 Secondary Endpoints

- Safety and Tolerability Variables:
  - Adverse Events (AEs)
  - Physical and neurological examination findings
  - Vital signs (BP and HR),
  - o 12-lead ECG (HR, PR, QRS, QTcB, QTcF), will be analysed ad hoc for safety and for the final data base and report by central reading
  - Clinical laboratory tests
    - Haematology: haemoglobin, haematocrit, mean corpuscular volume (MCV), mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC), platelets, reticulocytes, white blood cells (WBC) including differential, red blood cells (RBC);
    - Coagulation: activated partial thromboplastin time (aPTT), prothrombin time (PT);
    - Biochemistry: serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (AP), gamma-glutamyl transpeptidase (GGT), lactate dehydrogenase (LDH), creatine kinase (CK), amylase, lipase, glucose, cholesterol (HDL, LDL, total), triglycerides, creatinine, urea, uric acid, bilirubin (total and conjugated), total protein, sodium, potassium, calcium, chloride and magnesium;
    - Urinalysis: by dipstick glucose, ketone bodies, specific gravity, occult blood, pH, proteins, leucocytes, bilirubin, urobilinogen, nitrites, and microscopy (reflex).

### 4.2.3 Exploratory Endpoints

- Pharmacokinetic:
  - o AUC<sub>0-7d,norm</sub>, C<sub>max,norm</sub>, t<sub>1/2,0-24h</sub>, t<sub>1/2,0-7d</sub>, t<sub>max</sub>, MRT, points terminal

### 4.3 Statistical Hypotheses

Except for the analysis of pharmacokinetic data, no formal statistical testing will be done.

# 5 Study Design

This is a single-centre, open-label, randomized, parallel-group relative bioavailability study in healthy men. The study will be done in 2 parts, as follows:

- Part 1 single oral doses of 5 mg emodepside will be tested:
  - Part 1a the LSF (reference formulation) and 2 new IR-tablet formulations (test formulations) will be administered in the fasted state.
  - Part 1b the 2 new IR-tablet formulations will be administered in the fed state (high-fat, high-calorie meal).
- Part 2 single oral doses of 10 mg (2 x 5 mg) emodepside will be tested: depending on the results from Part 1, one or both IR-tablet formulations will be administered in the fasted state.

The treatments in each study part are summarised in Table 1.

Table 1. Planned treatments by dose, formulation and condition

| Part | Treatment | Formulation, dose and condition | Number of subjects |
|---|---|---|---|
| Part 1a | A | 5 mg emodepside LSF, fasted | 12 |
| | В | 5 mg emodepside IR-tablet #406, fasted | 12 |
| | C | 5 mg emodepside IR-tablet #416, fasted | 12 |
| Part 1b | D | 5 mg emodepside IR-tablet #406, fed | 12 |
| | E | 5 mg emodepside IR-tablet #416, fed | 12 |
| Part 2 | F* | 2 x 5 mg emodepside IR-tablet #406, fasted | 12 |
| | G* | 2 x 5 mg emodepside IR-tablet #416, fasted | 12 |

<sup>\*</sup> one or both treatments may be tested, depending on results from Part 1

Up to 84 healthy volunteers will be enrolled, in up to 7 treatment arms made up of 12 subjects each.

The 36 subjects in Part 1a will be randomised to one of 3 treatments (A, B or C). The 24 subjects in Part 1b will be randomised to one of 2 treatments (D or E). Parts 1a and 1b may proceed in parallel, or may be done sequentially.

After at least 10 subjects in each arm have received treatment in Part 1, and data up to 72 h after dosing are available, there will be a Dose Decision Meeting to determine which treatment(s) will be tested in Part 2 (see section 7.5).

In Part 2, either treatment F, G or both F and G will be tested. There will be 12 subjects enrolled for each treatment tested. If both treatments are tested, they will be done in parallel, and subjects will be randomised to one of the 2 treatments.

The study will be performed in a single site specialized in Phase 1 studies.

HMR code: 17-008

Sponsor code: DNDI-EMO-03

### **6** Time and Events Table

| | Screening | Inpatient | | | | | | | Follow-up | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day -28 to -2 | Day -1 | | | | | | | Day 0 | ) | | | | | | Da | y 1 | Day 2 | Day 3 | Day 5 | Day 7 |
| | | hours | -1 | 0 | 0.25 | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 6 | 8 | 12 | 24 | 36 | 48 | 72 | 120 | 168 |
| Subject demographics and informed consent | X | | | | | | | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria -<br>Eligibility check | X | Х | | | | | | | | | | | | | | | | | | | |
| Medical history/prior medication | X | | | | | | | | | | | | | | | | | | | | |
| Inpatient stay | | < | | | | | | | | | | | | | | | | | | | |
| Administration of emodepside <sup>1</sup> | | | | Х | | | | | | | | | | | | | | | | | |
| Outpatient visit | Х | | | | | | | | | | | | | | | | | | | Х | Х |
| Drugs of abuse screen | X | Х | | | | | | | | | | | | | | | | | | | |
| Alcohol breath test | X | Х | | | | | | | | | | | | | | | | | | | |
| Physical and neurological examination <sup>2</sup> | х | Х | | | | | | | Х | | | | | | | Х | Х | Х | Х | Х | х |
| Vital signs <sup>3</sup> | Х | | Х | | | Х | Х | Х | Х | | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х |
| 12-lead safety ECG <sup>4</sup> | Х | | Х | | | Χ | Х | Χ | Х | | Х | Х | | Х | Х | Х | | Х | Χ | Х | Х |
| Laboratory safety tests <sup>5,6</sup> | X | | Х | | | | | | | | | | | | | Х | | Х | Χ | Х | Х |
| Serology <sup>7</sup> | Х | | | | | | | | | | | | | | | | | | | | |
| Blood samples for assay of emodepside <sup>6</sup> | | | Х | | х | Х | Х | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х |
| AE questioning <sup>8</sup> | <u> </u> | | | | | • | | | | | | | | | | | | | | | $\overline{\rightarrow}$ |

- 1. Subjects in Part 1a and Part 2 will fast for 10 h before until at least 4 h after dosing. Subjects in Part 1b will be given a high-calorie, high-fat breakfast approximately 30 min before dosing, which they must finish at least 5 min before dosing. Standard meals will be served at approximately 5 h (lunch), 8 h (snack) and 12 h (dinner) after dosing on Day 0. Procedures scheduled at the same time as a meal will be completed before the meal.
- 2. A full physical examination will be done at Screening and Follow-up. A brief (symptom-directed) physical examination and short neurological examination will be undertaken at all other time points. Any abnormalities will trigger a full neurological examination and/or opening of an AE as appropriate. Height, weight and body mass index (BMI) will be assessed at screening, and weight will be assessed on Day –1.
- 3. Vital signs will comprise supine blood pressure and heart rate. Subjects should rest in the supine position for at least 10 min before vital signs measurements. Vital signs will be measured in triplicate at screening and pre-dose (-1 h); single measurements at all other time points. Body temperature will be measured on day -1.

HMR code: 17-008

Sponsor code: DNDI-EMO-03

4. Subjects should rest in the supine position for 10 min before ECG measurements. Measurement in triplicate at screening and pre-dose (-1 h); single measurements all other time points.

- 5. Blood and urine samples for clinical laboratory safety tests (haematology, biochemistry, coagulation and urinalysis).
- 6. Subjects should rest in the supine position for 10 minutes before blood is drawn (if possible).
- 7. Serology tests will comprise HIV 1 & 2 and hepatitis B & C.
- 8. Adverse event monitoring will be done throughout the study, but scheduled questioning will be done at the time points of scheduled blood draws.

# 7 Planned Analyses

# 7.1 Interim Analyses

The decision to go ahead with one or both treatments in Part 2 (10mg [2 x 5mg] of IMP) will be made based on the safety, tolerability and PK of the treatments in Part 1 (5mg of IMP).

The dose decision will be made by the Safety Review Group (SRG) at the Safety Review Meeting. The treatments will not be decided until the SRG has reviewed the safety, tolerability and PK data of at least 10 subjects per treatment. Safety, tolerability and PK data up to a minimum of 72 h post-dose should be reviewed before a decision can be made.

#### 7.1.1 Persons responsible for analysis

Toni Mitchell (HMR) Statistician

Nick Jackson (HMR) SAS Programmer

# 7.2 Final Analysis

Each part of the study (Part 1 and Part 2) will have a separate database and will be analysed and reported separately. Each database will be locked once all subjects have completed, data have been entered, all queries resolved and protocol deviations identified for that part of the study. Final analyses will be carried out following database lock for each individual part of the study.

#### 7.2.1 Persons responsible for analysis

Helen Topping (HMR) Statistician

Nick Jackson (HMR) SAS Programmer

Duyen Unsworth (HMR) Data Manager

# 8 Sample Size Considerations

# 8.1 Sample Size Assumptions

No formal statistical sample size estimation has been performed, due to the exploratory nature of this study.

10 subjects per treatment arm is considered sufficient to examine the safety and tolerability of emodepside, as well as the PK after single doses. However, 12 subjects will be recruited and enrolled per treatment arm to ensure a minimum of 10 evaluable subjects complete the study.

# 9 Analysis Populations

The following populations will be identified:

Safety Population: All subjects who received at least one dose of IMP.

PK Concentration Population: All subjects who received at least one dose of IMP and

for whom a PK sample has been analysed.

PK Parameter Population: All subjects in the PK Concentration Population for

whom PK parameters can be derived.

In all populations, treatment will be assigned based upon the treatment subjects actually received, regardless of the treatment to which they were randomized.

The primary endpoint will be analysed using the PK Parameter population.

# 9.1 Analysis Datasets

All analysis datasets will be based on observed data, except as outlined in Section 12.2.

# 10 Treatment Comparisons

The treatment comparison of interest is test (IR-tablet formulations) versus reference (LSF).

# 11 General Considerations for Data Analyses

### 11.1 Data Display Treatment and Other Subgroup Descriptors

The sort order for treatment groups will be treatment in ascending dose order. When a total column is included, it immediately follows the treatment groups which it aggregates.

Listings of data will be sorted and displayed by treatment group, subject number, and also by date and time if applicable.

The treatment descriptions to be used on all tables and listings are:

| Short Description |
|------------------------|
| LSF 5 mg [fasted] |
| IR #406 5 mg [fasted] |
| IR #416 5 mg [fasted] |
| IR #406 5 mg [fed] |
| IR #416 5 mg [fed] |
| IR #406 10 mg [fasted] |
| IR #416 10 mg [fasted] |

# 11.2 Conventions for Summary Statistics and Data Displays

The minimum set of summary statistics for numeric variables will be: n, mean, standard deviation (or standard error), median, minimum, and maximum. 95% confidence intervals will be presented where appropriate for data interpretation.

Categorical data will be summarised in frequency tables with n and percentage. Summaries of a categorical variable will include all recorded values.

The minimum and maximum values will be presented with the same number of decimal places as the raw data collected on the CRF (or to 3 significant figures for derived parameters less than 100 and as integers for values more than 99). The mean and percentiles (e.g. median, Q1, and Q3) will be presented using one additional decimal place. The standard deviation and standard error will be presented using two additional decimal places.

# 12 Data Handling Conventions

### 12.1 Premature Withdrawal and Missing Data

All subjects who withdraw prematurely from the study and received the study drug will be included in the statistical analyses.

If a subject completes the treatment period but has missing data, then this will be made apparent in the subject listings. Missing data will not be imputed except for as outlined in Section 12.2.

If the study is prematurely discontinued, all available data will be listed and a review will be carried out to assess which statistical analyses are still considered appropriate.

Data collected at unscheduled time points during the study will not be used in the summaries or data analyses. They will be included in the listings.

If time information (i.e. hours and/or minutes) for adverse events or concomitant medication is missing, but the day is present, then the time will be calculated in days. If date information is partial or missing, then any derived times (e.g. AE start time from last study medication) will be listed as missing.

Conventions for handling missing plasma concentrations are given in Appendix B.

#### 12.2 Derived and Transformed Data

Baseline will be considered to be the latest value obtained before study drug administration (e.g. Day 0, pre-dose; or Day -1 if not recorded pre-dose; or Screening if not recorded elsewhere (e.g. body weight)).

Laboratory data will be reported in standard units. Out-of-range laboratory tests may be repeated. If a test is out-of-range at a baseline time point and repeated before dosing, the latest repeat value before dosing will be used as baseline. However, if a test is out-of-range and repeated at any other time during the study, the out-of-range value (not the repeat value) will be included in statistical summaries.

Triplicate ECG and vital sign measurements will be made at pre-dose on Day 0 and the mean of the three measurements for each subject will be used as their baseline value for that session.

The pharmacokinetic parameters to be derived are given in Appendix B.

#### 12.3 Assessment Windows

No assessment windows are defined for this report.

### 12.4 Values of Potential Clinical Importance

Any laboratory value outside the reference interval for that variable will be flagged with an 'H' if it is higher than the reference interval, and with an 'L' if it is lower. Additionally, if, during the course of the trial, a variable changes from baseline (Day 0 pre-dose) by more than a predetermined amount (as defined by the Principal Investigator, Appendix A), that value will receive a flag 'I' if increased, or 'D' if decreased. Therefore, if a value both falls outside the reference interval and alters from the baseline value by more than the predetermined amount, it will attract a double flag and will be considered to be potentially clinically important.

A vital signs result will be considered to be of potential clinical importance if it falls outside the relevant range below:

| Vital Sign | Range |
|------------------------------------------------|------------------|
| Supine/semi-recumbent systolic blood pressure | 85–160 mm Hg |
| Supine/semi-recumbent diastolic blood pressure | 40–90 mm Hg |
| Supine/semi-recumbent heart rate | 35-100 beats/min |
| Respiration rate | 8–20 per min |
| Oral temperature | 35.5–37.8°C |

QT, QTcB or QTcF > 450 msec and increases in QT, QTcB or QTcF from baseline (Day 1 pre-dose) of > 30 msec will be considered to be potentially clinically important.

# 13 Study Population

### 13.1 Disposition of Subjects

The disposition of all subjects in the safety population will be summarized including: number of subjects randomized (or treated, for non-randomised groups); number completing the study, by treatment; and number discontinued from the study. The number of subject in each analysis population will be summarized by treatment.

All subjects who withdraw or are withdrawn from the study will be listed, by treatment, with the reason for withdrawal.

A listing of analysis populations will be provided.

#### 13.2 Protocol Deviations

Before closing the database, data listings will be reviewed to identify any significant deviations and determine whether the data should be excluded from any analysis populations.

Major protocol deviations include subjects who:

- Entered the study even though they did not satisfy the entry criteria.
- Met the criteria for withdrawal from the study but were not withdrawn.
- Received the wrong treatment or incorrect dose.
- Received an excluded concomitant therapy.
- Received investigational product(s) past the expiration date.

In addition, subjects with minor time deviations (measurements taken outside the allowable windows) will be identified. Allowable time windows for pharmacokinetic samples and other procedures are given in section 8.8 of the study protocol.

### 13.3 Demographic and Baseline Characteristics

Demographic and baseline characteristics (e.g. physical examination, vital signs and ECGs) will be listed and summarised.

Subjects who take concomitant medication will be listed. All non-trial medication will be coded using the version of the WHODrug Global that is current when the database is locked.

### 13.4 Treatment Compliance

Dates and times of dosing will be listed.

# 14 Safety Analyses

Summaries and listings of safety data will use the safety population.

### 14.1 Extent of Exposure

The dates and times of treatment dosing will be listed to indicate exposure to the study medication

#### 14.2 Adverse Events

Adverse events will be coded using the version of the Medical Dictionary for Regulatory Activities (MedDRA) which is current at the time of database lock (version 20.1 or higher).

All adverse events will be listed

The number of subjects with at least one treatment-emergent adverse event (TEAE) will be tabulated by actual treatment and MedDRA system organ class. A treatment-emergent adverse event is defined as an event emerging during treatment having been absent pretreatment or having worsened relative to pre-treatment<sup>1</sup>.

For each of the following, the number of adverse events and the number of subjects with adverse events will be summarised:

- TEAEs by system organ class and preferred term
- TEAEs by system organ class, preferred term and severity
- Drug-related ("Related" as recorded by the Investigator) TEAEs by system organ class and preferred term

Subjects with more than one TEAE will be counted only once, at the greatest severity or causality, for each system organ class/preferred term. Multiple TEAEs in a subject will be counted once per system organ class and preferred term. Adverse events with missing severity and/or causality will be treated as severe and related, respectively.

Summaries will be sorted by system organ class and decreasing total incidence of preferred term.

# 14.3 Deaths, Serious Adverse Events and Other Significant Adverse Events

Deaths and serious adverse events will be listed separately (fatal events separate from non-fatal events). Other significant adverse events, as identified by the investigator in the CRF, will be listed separately.

### 14.4 Adverse Events Leading to Withdrawal from the Study

Adverse events leading to withdrawal will be listed separately.

### 14.5 Clinical Laboratory Evaluations

Data from haematology, coagulation, clinical chemistry and urinalysis will be summarised by treatment.

Urinalysis parameters will also be listed

All laboratory values of potential clinical importance will be listed and all related laboratory results (i.e. haematology or clinical chemistry) for subjects with values of potential clinical importance will be listed, separately. Frequencies of laboratory values of potential clinical importance will be summarised.

### 14.6 Other Safety Measures

#### 14.6.1 Vital signs

Vital signs evaluation at each planned assessment, and change in vital signs from baseline (Day 0 pre-dose in the current treatment period) at each planned post-baseline assessment (with or without potential clinical significance) will be summarised by actual treatment.

Vital signs data of potential clinical importance will be listed.

#### 14.6.2 ECG

QT interval data will be presented using Bazett's (QTcB) and Fridericia's (QTcF) corrections.

ECG data will be summarised by treatment and time point. Differences from baseline (Day 0 pre-dose) will be summarised by treatment and time point.

The number of subjects with a potentially clinically important ECG value will be summarised by actual treatment and time point, giving the numbers of subjects with QT, QTcB or QTcF > 450 msec, > 480 msec and > 500 msec, and the numbers of subjects with increases in QT, QTcB or QTcF from baseline of > 30 msec and > 60 msec<sup>3</sup>. A supporting listing of all subjects with an ECG value of potential clinical importance and a separate listing of ECG findings classified as abnormal by the Investigator will also be provided.

#### 14.6.3 Physical and neurological examination

Abnormal physical and neurological examination findings will be listed.

# 15 Pharmacokinetic Analyses

Analytical Services International Ltd, London, U.K will measure the plasma concentrations of emodepside. The pharmacokinetic analysis will be done by HMR. Pharmacokinetic parameters will be calculated using WinNonlin, version 7 or higher.

The pharmacokinetic parameters to be derived are given in Appendix B.

PK Concentration data will be summarised using the PK concentration population. PK parameters will be summarised using the PK Parameter population.

For log normally distributed parameters, the primary measure of central tendency will be the geometric mean<sup>4</sup>; for other parameters, it will be the arithmetic mean or median.

For all variables N (number of subjects receiving the treatment/formulation in the population), n (number of observations), arithmetic mean, median, minimum, maximum, SD, %CV, and the 95% confidence interval for the arithmetic mean will be provided. For log-transformed variables, all of the above plus the geometric mean, which is the anti-logged arithmetic mean of log-transformed variables, its 95% confidence interval and the SD of the logs will be provided.

The between-subject CV will be calculated using:

- 1. %CVb = 100 \* (SD/Mean) with SD and Mean of untransformed data
- 2. %CVb =  $100 * \sqrt{(\exp(SD)^2 1)}$  with SD of log-transformed data

### 15.1 Pharmacokinetic Concentration Data

The plasma concentrations will be listed and summarised by treatment. Individual and mean plasma concentration—time profiles will be presented graphically.

#### 15.2 Pharmacokinetic Parameters

The pharmacokinetic parameters will be listed and summarised by treatment.

To assess the relative bioavailability, analysis of variance (ANOVA) models will be fitted to the tablet (test) and solution (reference) data with the logarithm of the pharmacokinetic parameters  $AUC_{0-7d}/Dose$  or  $C_{max}/Dose$  as the dependent variable, and formulation as a fixed effect. The point estimates least squares (LS)-means and 90% confidence intervals for the ratios "B/A" and "C/A" will be calculated in Part 1a. In Part 2, "F/A" and/or "G/A" will be calculated. The acceptance range 80 - 125% will be applied for these assessments.

In part 1, to assess the effect of food, ANOVA models will be fitted to the data with the logarithm of the pharmacokinetic parameters  $AUC_{0-7d}/Dose$  or  $C_{max}/Dose$  as the dependent variable, and fed (test) or fasted (reference) as a fixed effect. The point estimates and 90% confidence intervals for the ratios "D/B" and "E/C" will be calculated. The acceptance range 80-125% will be applied for the assessment of a potential food effect.

To assess dose proportionality, for each tablet type, exploratory ANOVA models will be fitted to the relevant fasted data in Parts 1 and 2 with the logarithm of the pharmacokinetic parameters  $AUC_{0-7d}$  or  $C_{max}$  as the dependent variable and dose as a fixed effect. The ratios "F/B" and/or "G/C" will be calculated, with their 95% confidence interval.

#### 16 References

- 1. International Conference on Harmonization, 1998. Statistical Principles for Clinical Trials ICH Harmonised Tripartite Guideline. Guidance for Industry, E9, FDA federal register, Vol 63, 1998, p49583. Available at: http://www.fda.gov/cder/guidance.
- 2. International Conference on Harmonization, 1995. Structure and Content of Clinical Study Reports ICH Harmonised Tripartite Guideline. Guidance for Industry, E3, FDA federal register, Vol 61, 1996, p37320. Available at: http://www.fda.gov/cder/guidance.
- 3. International Conference on Harmonisation, 2005. Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs. Concept paper, Guidance for Industry, E14, Center for Drug Evaluation and Research (CDER). Available at: http://www.fda.gov/cder/guidance/6922fnl.htm.
- 4. Julious, SA & Debarnot, CAM (2000) "Why are Pharmacokinetic Data Summarised by Arithmetic Means?", Journal of Biopharmaceutical Statistics, 10 (1), p55-71

### 17 ATTACHMENTS

# 17.1 Table of Contents for Data Display Specifications

For overall page layout refer to Appendix C.

Tables, figures and listings will be labelled A (for Part 1) and B (for Part 2), e.g. 14.1A, 14.1B. Separate tables will be produced for Parts A and B.

The numbering in the tables below will take precedence over the numbering in the shells.

The following tables and figures will be produced (templates provided in Section 17.2.1 and 17.2.2):

| Table | Description | Population | Source<br>Listing | Template (Shells below) |
|---|---|---|---|---|
| 10.1 | Summary of Subject Disposition | Safety | 16.2.1.2,<br>16.2.3.1 | T_SD1 |
| 14.1 | DEMOGRAPHIC DATA | | | |
| 14.1 | Summary of Demographic Characteristics | Safety | 16.2.4.1 | <u>T_DM1</u> |
| 14.2 | PHARMACOKINETIC AND PHARMACODYNAMIC DATA | | | |
| 14.2.1 | Summary of Emodepside Plasma Pharmacokinetic Concentration-<br>Time Data (ng/mL) | PK Concentration | 16.2.6.1 | <u>T_PK1</u> |
| 14.2.2 | Summary of Derived Emodepside Plasma Pharmacokinetic Parameters | PK Parameter | 16.2.6.2 | <u>T_PK3</u> |
| 14.2.3 | Summary of Log-Transformed Derived Emodepside Plasma<br>Pharmacokinetic Parameters | PK Parameter | 16.2.6.2 | <u>T_PK4</u> |
| 14.2.4 | Summary of Relative Bioavailability of Emodepside | PK Parameter | 16.2.6.2 | <u>T_PK6</u> |
| 14.2.5 | Assessment of the Effect of Food on the PK of Emodepside | PK Parameter | 16.2.6.2 | <u>T_PK6</u> |
| 14.2.6 | Summary of Dose Proportionality Analysis of Emodepside | PK Parameter | 16.2.6.2 | <u>T_PK8</u> |
| 14.3 | SAFETY DATA | | | |
| 14.3.1.1 | Summary of Treatment-Emergent Adverse Events | Safety | 16.2.7.1 | <u>T_AE1</u> |
| 14.3.1.2 | Summary of Treatment-Emergent Adverse Events by Severity | Safety | 16.2.7.1 | <u>T_AE1</u> |
| 14.3.1.3 | Summary of Drug-Related Treatment-Emergent Adverse Events | Safety | 16.2.7.1 | <u>T_AE1</u> |
| 14.3.2.1 | Listing of Fatal Adverse Events | Safety | 16.2.7.1 | L_AE1_PG |
| 14.3.2.2 | Listing of Non-Fatal Serious Adverse Events | Safety | 16.2.7.1 | L_AE1_PG |
| 14.3.2.3 | Listing of Other Significant Adverse Events | Safety | 16.2.7.1 | L_AE1_PG |
| 14.3.3 | Narratives of deaths, other serious and significant adverse events | Safety | | - |
| 14.3.4 | Summary of Laboratory Values of Potential Clinical Importance | Safety | 16.2.8.1<br>16.2.8.3 | <u>T_LB1</u> |
| 14.3.5.1 | Summary of Chemistry Laboratory Values | Safety | 16.4 | <u>T_LB2</u> |
| 14.3.5.2 | Summary of Haematology Laboratory Values | Safety | 16.4 | <u>T_LB2</u> |
| 14.3.5.3 | Summary of Coagulation Values | Safety | 16.4 | <u>T_LB2</u> |
| 14.3.5.4 | Summary of Urinalysis Dipstick Results | Safety | 16.2.8.5 | T_UR1 |
| 14.3.6 | Summary of Vital Signs | Safety | 16.4 | <u>T_VS1</u> |
| 14.3.7.1 | Summary of ECG Values | Safety | 16.4 | T_EG2 |

| Table | Description | Population | Source<br>Listing | Template (Shells below) |
|---|---|---|---|---|
| 14.3.7.2 | Summary of ECG Values and Changes in ECG Values of Potential | Safety | 16.2.9.2 | T EG3 |
| | Clinical Importance | | | |

| Figure | Description | Population | Source<br>Listing | Template (Shells below) |
|---|---|---|---|---|
| 14.3 | PHARMACOKINETIC AND PHARMACODYNAMIC DATA | | | |
| 14.2.1 | Individual Emodepside Plasma Concentration-Time Plots (Linear and | PK | 16.2.6.1 | E DV1 |
| 14.2.1 | Semi-log) | Concentration | 10.2.0.1 | <u>F_PK1</u> |
| 14.2.2 | Geometric mean (+/- SD) Emodepside Plasma Concentration-Time | PK | 16.2.6.1 | F PK2 |
| 14.2.2 | Plots (Linear and Semi-log) | Concentration | 10.2.0.1 | <u>r_rkz</u> |
| 14.3 | SAFETY DATA | | | |
| 14.3.1 | Individual Systolic Blood Pressure-Time Plots | Safety | 16.4 | F SAF1 |
| 14.3.2 | Individual Diastolic Blood Pressure-Time Plots | Safety | 16.4 | F_SAF1 |
| 14.3.3 | Individual Heart Rate-Time Plots | Safety | 16.4 | F SAF1 |
| 14.3.4 | Individual QTcF-Time Plots | Safety | 16.4 | F SAF1 |
| 14.3.5 | Individual QTcB-Time Plots | Safety | 16.4 | F SAF1 |

The following abbreviated listings will be produced (templates provided in Section 17.2.3):

| Listing | Description | Template<br>(Shells below) |
|---|---|---|
| 16.2.1 | Study dates & disposition of subjects | |
| 16.2.1.1 | Listing of Study Dates | L SD1 PG |
| 16.2.1.2 | Listing of Reasons for Withdrawal | L SD2 PG |

| Listing | Description | Template<br>(Shells below) |
|---|---|---|
| 16.2.2 | Protocol deviations | (Shens below) |
| 16.2.2.1 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | L DV1 PG |
| 16.2.2.2 | Listing of Subjects with Time Deviations | L TD1 PG |
| 16.2.2.3 | Listing of Subjects with Other Protocol Deviations | L DV2 PG |
| 16.2.3 | Analysis sets, including subjects excluded from analysis | |
| 16.2.3.1 | Listing of Analysis Populations | L AN1 PG |
| 16.2.4 | Demographic data & concomitant medication | |
| 16.2.4.1 | Listing of Demographic Characteristics | L DM1_PG |
| 16.2.4.2 | Listing of Concomitant Medications | L_CM1_PG |
| 16.2.5 | Study drug administration | |
| 16.2.5.1 | Listing of Exposure Data | L EX1 PG |
| 16.2.6 | Pharmacokinetic and pharmacodynamic data | |
| 16.2.6.1 | Listing of Emodepside Plasma Pharmacokinetic Concentration-Time Data | L PK1 PG |
| 16.2.6.2 | Listing of Derived Emodepside Plasma Pharmacokinetic Parameters | L PK4 PG |
| 16.2.6.3 | Individual Emodepside Plasma Concentration-Time Plots (log scale) for Estimation of | <u>F_PK10</u> |
| <b>-</b> | λz, with Regression Line | |
| 16.2.7 | Adverse events | |
| 16.2.7.1 | Listing of All Adverse Events | L AE1 PG |
| 16.2.7.2 | Listing of Serious Adverse Events | L_AE1_PG |
| 16.2.7.3 | Listing of Adverse Events Leading to Withdrawal from Study | L AE1 PG |
| 16.2.8 | Laboratory values | |
| 16.2.8.1 | Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance | L LB1 PG |
| 16.2.8.2 | Listing of All Clinical Chemistry Laboratory Data for Subjects with PCI Abnormalities* | L_LB2_PG |
| 16.2.8.3 | Listing of Haematology Abnormalities of Potential Clinical Importance | L LB1 PG |
| 16.2.8.4 | Listing of All Haematology Laboratory Data for Subjects with PCI Abnormalities* | L_LB2_PG |
| 16.2.8.5 | Listing of Urinalysis Data | <u>L_URI_PG</u> |
| 16.2.9 | Vital signs, ECG variables, physical and neurological findings | |
| 16.2.9.1 | Listing of Vital Signs of Potential Clinical Importance | L_VS1_PG |
| 16.2.9.2 | Listing of ECG Values of Potential Clinical Importance | L_EG1_PG |

ListingDescriptionTemplate<br/>(Shells below)16.2.9.3Listing of Abnormal ECG FindingsL EG2 PG16.2.9.4Listing of Abnormal Physical Examination FindingsL PE1 PG16.2.9.5Listing of Abnormal Neurological Examination FindingsL NE1 PG

Complete listings of all data collected in this study will also be produced.

<sup>\*</sup> ICH does not require full listings of lab data so only subjects with double-flagged values will be listed.

# 17.2 Data Display Specifications

### 17.2.1 Table Outlines

#### Template T\_SD1

Table 10.1 Summary of Subject Disposition

| Population | Status | Reason for Withdrawal | Treatment 1 | Treatment 2 | Etc | All Subjects |
|---|---|---|---|---|---|---|
| | | | n (%) | n (%) | | n (%) |
| Safety | Included | | XX | XX | | XX |
| | Completed | | xx (xx) | xx(xx) | | xx (xx) |
| | Withdrawn | | | | | |
| | | Death | xx (xx) | xx(xx) | | xx (xx) |
| | | Adverse Events | xx (xx) | xx(xx) | | xx (xx) |
| | | Withdrawal by subject | xx (xx) | xx(xx) | | xx (xx) |
| | | Physician decision | xx (xx) | xx (xx) | | xx(xx) |
| | | Protocol violation | xx (xx) | xx(xx) | | xx (xx) |
| | | Pregnancy | xx (xx) | xx(xx) | | xx (xx) |
| | | Study terminated by | xx (xx) | xx(xx) | | xx (xx) |
| | | Sponsor | | | | |
| | | Lost to follow-up | | | | |
| | | Other | xx (xx) | xx (xx) | | xx (xx) |
| Alternative 1 (if applicable) | Included | | xx (xx) | xx (xx) | | xx (xx) |
| Alternative 2 (if applicable) | Included | | xx (xx) | xx (xx) | | xx (xx) |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups

### Template T\_DM1

Table 14.1 Summary of Demographic Characteristics

| Variable | Statistics | Treatment 1 | Treatment 2 | Etc | All Subjects (N=xx) |
|---|---|---|---|---|---|
| | | (N=xx) | (N=xx) | | |
| Age (y) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Min | | | | |
| | Max | | | | |
| Gender | n | | | | |
| | Female | | | | |
| | Male | | | | |
| Race | American Indian or Alaskan | | | | |
| | Native | | | | |
| | Asian | | | | |
| | Black | | | | |
| | Native Hawaiian or other | | | | |
| | Pacific Islander | | | | |
| | White | | | | |
| | Other | | | | |
| Ethnicity | Hispanic or Latino | | | | |
| | Not Hispanic or Latino | | | | |
| Height (cm) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Min | | | | |
| | Max | | | | |
| Weight (kg) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |

| Variable | Statistics | Treatment 1 | Treatment 2 | Etc | All Subjects (N=xx |
|---|---|---|---|---|---|
| | | (N=xx) | (N=xx) | | |
| | Min | | | | |
| | Max | | | | |
| BMI (kg/m2) | n | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Min | | | | |
| | Max | | | | |
| Smoker | n | | | | |
| | % | | | | |
| Cigarettes* | n | | | | |
| (daily) | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Min | | | | |
| | Max | | | | |
| Alcohol* | n | | | | |
| (units/week) | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Min | | | | |
| | Max | | | | |
| Xanthine* | n | | | | |
| (units/week) | | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | Min | | | | |
| | Max | | | | |

<sup>\*</sup>includes only those subjects who smoke/drink alcohol/drink beverages containing xanthine

Source: Listing 16.2.xx

HMR code: 17-008

Sponsor code: DNDI-EMO-03

Programming notes: Continued with all treatment groups and additional demographic characteristics

#### Template T\_PK1

Table 14..2.xx Summary of Emodepside Plasma Pharmacokinetic Concentration-Time Data [units]

| Treatment<br>(N=xx) | Planned<br>Relative<br>Time | n | No.<br>Imputed | Mean | 95% CI | SD | %CVb | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment 1 | 1h | | · | | | | | | | |
| (N=xx) | | | | | | | | | | |
| Treatment 2 | | | | | | | | | | |
| (N=xx) | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels and timepoints

Means, SD, CI and CV should only be calculated if ≥2/3 individual values are >LLOQ

#### Template T\_PK3

Table 14..2.xx Summary of Derived Emodepside Plasma Pharmacokinetic Parameters

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels and parameters

HMR code: 17-008

Sponsor code: DNDI-EMO-03

#### Template T\_PK4

Table 14..2.xx Summary of Log-Transformed Derived Emodepside Plasma Pharmacokinetic Parameters

| Parameter | Treatment (N=xx) | n | Geom Mean | 95% CI | SD (logs) | %CVb |
|---|---|---|---|---|---|---|
| AUC <sub>last</sub> (units) | | | | | | |
| C <sub>max</sub> (units) | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels and parameters

#### Template T\_PK6

Table 14.2.xx Summary of Relative Bioavailability of Emodepside

| | | | L | SMeans | Test vs | Reference |
|---|---|---|---|---|---|---|
| Parameter | Test Formulation Reference Tes | | Test | Ref | Ratio (%) | 90% CI |
| C <sub>max/</sub> Dose<br>(units) | #406 5 mg | LSF | xx.x | xx.x | xxxx.x | xxxx.x, xxxx.x |
| | #416 5 mg | | XX.X | xx.x | xxxx.x | xxxx.x, xxxx.x |
| AUC <sub>0-7d/</sub> Dose<br>(units) | #406 5 mg | LSF | xx.x | xx.x | xxxx.x | xxxx.x, xxxx.x |
| . , | #416 5 mg | | XX.X | XX.X | xxxx.x | xxxx.x, xxxx.x |

Source: Listing 16.2.xx

Programming notes: For bioavailability In part 1a calculate values for "B/A" and "C/A"

In part 2 calculate values for "F/A" and "G/A"

For food effect calculate for part 1 only values for "D/B" and "E/C"

Sponsor code: DNDI-EMO-03

### Template T\_PK8

Table 14.2.xx Summary of Dose Proportionality Analysis of Emodepside

| | | 10mg vs 5 | 5 mg |
|-------------|-----------------------------|-----------|----------------|
| Formulation | Parameter | Ratio (%) | 95% CI |
| #406 5 mg | C <sub>max</sub> (units) | xxxx.x | xxxx.x, xxxx.x |
| | AUC <sub>0-7d</sub> (units) | xxxx.x | xxxx.x, xxxx.x |

Source: Listing 16.2.xx

Programming notes: Continue with all formulations. Calculate "F/B" and/or "G/C"

HMR code: 17-008

Sponsor code: DNDI-EMO-03

#### Template T\_AE1

Table 14.3.3.xx Summary of Treatment-Emergent Adverse Events

| | | Treatment 1 (N=xx) | Treatment 2 (N=xx) Etc |
|---|---|---|---|
| System Organ Class | Preferred Term | n (%) | n (%) |
| Number of subjects with AEs | | x (xx.x) | x (xx.x) |
| Gastrointestinal disorders | Total number of subjects | x (xx.x) | x (xx.x) |
| | Abdominal discomfort | x (xx.x) [xx] | x (xx.x) [xx] |
| | Abdominal pain | x (xx.x) [xx] | x (xx.x) [xx] |
| | $\downarrow$ | | |
| Nervous system disorders | Total number of subjects | | |
| | Dizziness | | |
| | Headache | | |
| | $\downarrow$ | | |
| $\downarrow$ | $\downarrow$ | | |

n = number of subjects (subjects with ≥1 adverse event are counted only once per system organ class and preferred term

[] = number of adverse events Based on MedDRA version xx.x

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups

SOCs and PTs are sorted in decreasing order of frequency

Presented for all applicable MedDRA system organ classes and terms.

HMR code: 17-008

Sponsor code: DNDI-EMO-03

#### Template T\_LB1

Table 14.3.4.xx Summary of Laboratory Values of Potential Clinical Importance

| | | Planned Relative | | Doub | le Flags |
|---|---|---|---|---|---|
| Laboratory Test (units) | Treatment | Time | n | HI | LD |
| | Treatment 1 (N=xx) | | | | |

H = Above reference interval, L = Below reference interval, I = Increase from baseline greater than pre-defined limit, D = Decrease from baseline greater than pre-defined limit

Source: Listing 16.2.xx

Programming notes: Continued with all tests, treatment groups and time points. n = total number of results for that parameter

#### Template T\_LB2

Table 14.3.5.xx Summary of Chemistry Laboratory Values

| | | | | | | Cha | ange f | rom Baselin | ie | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Test | | Planned | | | | | | | | | | | | |
| (units) | Treatment | Relative Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| | Treatment 1 (N=xx) | | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatments and time points
Sponsor code: DNDI-EMO-03

#### Template T\_UR1

Table 14.3.5.xx Summary of Urinalysis Dipstick Results

| | Planned Relative | e | Treatment 1 | L (N=xx) | Treatment 2 (N=xx | |
|---|---|---|---|---|---|---|
| Laboratory Test | Time | Result | n | % | n | % |
| | Time 1 | Positive | Х | х | | |
| | | Negative | Х | Χ | | |
| | | Not Done | x | | | |
| | Time 2 | Positive | | | | |
| | | Negative | | | | |
| | | Not Done | | | | |

Source: Listing 16.2.xx

Programming notes: Results recorded as received, e.g. Negative, Trace, etc; urine pH summarized as <5, 5-8, >8

Continued with all treatment groups and time points. The n's sum to N but the calculated percentages exclude Not Done.

#### Template T\_VS1

Table 14.3.6.xx Summary of Vital Signs

| | | | | | | | | | Chan | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Planned | | | | | | | | | | | |
| Variable (units) | Treatment | Relative Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median Min | Max |
| Systolic BP (mmHg) | Treatment 1 (N=xx) | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all variables, treatments and time points

Sponsor code: DNDI-EMO-03

### Template T\_EG2

Table 14.3.7.xx Summary of ECG Values

| | | | | | | | | | | Cl | hange | from Baseli | ne | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Planned Relative | | | | | | | | | | | | |
| Variable (units) | Treatment | Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Heart Rate (bpm) | Treatment 1 (N=xx) | | | | | | | | | | | | | |
| | Treatment 2 (N=xx) | | | | | | | | | | | | | |
| PR Interval (msec) | Treatment 1 (N=xx) | | | | | | | | | | | | | |
| | Treatment 2 (N=xx) | | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups and time points

Do not summarise RR or QRS axis

### Template T\_EG3

Table 14.3.7.xx Summary of ECG Values and Changes in ECG Values of Potential Clinical Importance

| | | Planned | | | | | | | >30-6 | 0 msec | >60 । | msec |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Relative | 451 – 48 | 30 msec | 481 – 5 | 00 msec | > 500 | ) msec | Incr | ease | Incr | ease |
| Variable | Treatment | Time | n | % | n | % | n | % | n | % | n | % |
| QT interval | Treatment 1 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | | Time 3 | | | | | | | | | | |
| | Treatment 2 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | | Time 3 | | | | | | | | | | |
| QTcB interval | Treatment 1 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | | Time 3 | | | | | | | | | | |
| | Treatment 2 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | | Time 3 | | | | | | | | | | |
| QTcF interval | Treatment 1 | Time 1 | | | | | | | | | | |
| | (N=xx) | Time 2 | | | | | | | | | | |
| | , , | Time 3 | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatments and time points. n = total number of results for that parameter

## 17.2.2 Figure Outlines

#### Template F\_PK1

Figure 16.2.4.xx Individual Emodepside Plasma Concentration-Time Plots (Linear and Semi-log)

Treatment x





Programming note: Plot will include all subjects for a given treatment group

#### Template F\_PK2

Figure 16.2.4.xx Geometric mean (+ SD) of Emodepside Plasma Concentration-Time Plots (Linear and Semi-log)



BLQ values are imputed to zero

Programming note: The SD is the geometric standard deviations

In Part 1, the following treatment comparisons will be plotted separately: LSF vs #406 5mg [fasted] and #416 5 mg [fasted], LSF vs #406 5 mg [fed] and #416 5 mg [fed], LSF vs #406 5mg [fed], LSF vs #416 5 mg [fed] and #416 5 mg [fed].

#### Template F\_PK10

Figure 16.2.xx Individual Emodepside Plasma Concentration-Time Plots (log scale) for Estimation of Lambda-z, with Regression Line



### Template F\_SAF1

Figure 14.3.1 Individual Systolic Blood Pressure-Time Plots



Programming note: Plots are by treatment groups
Continue with all parameters

Sponsor code: DNDI-EMO-03

## 17.2.3 Listing Outlines

Template L\_SD1\_PG

Listing 16.2.x.xx Listing of Study Dates

Treatment Subject Screening First dose Follow Up

Programming notes: Lists dates for screening, each dosing period and follow up

Template L\_SD2\_PG

Listing 16.2.x.xx Listing of Reasons for Withdrawal

Date of Study
Treatment Subject Withdrawal Day Reason

Programming notes: Reason for withdrawal is concatenation of reason and details

Template L\_DV1\_PG

Listing 16.2.x.xx Listing of Subjects with Inclusion/Exclusion Criteria Deviations

Treatment Subject Type Criterion

Exclusion

Sponsor code: DNDI-EMO-03

#### Template L\_TD1\_PG

Listing 16.2.x.xx Listing of Subjects with Time Deviations

| | | | Planned | | Allowed | Actual |
|-----|--------|---------|----------|-----------|-----------|-----------|
| | | | Relative | | deviation | deviation |
| Tre | atment | Subject | Time | Procedure | (h:min) | (h:min) |

Programming notes: Only include time deviations which exceed the allowed deviation

#### Template L\_DV2\_PG

Listing 16.2.x.xx Listing of Subjects with Other Protocol Deviations

Treatment Subject Protocol Deviation

### Template L\_AN1\_PG

Listing 16.2.x.xx Listing of Analysis Populations

Safety

Treatment Subject Population Population 1 Population 2 Etc.

## Template L\_DM1\_PG

Listing 16.2.x.xx Listing of Demographic Characteristics

| | | | | Age | | | | Height | Weight | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Date of visit | Date of birth | (y) | Gender | Race | Ethnic origin | (cm) | (kg) | BMI (kg/m2) | Etc (units) |
| Treatmen<br>↓ | t 1 | | | | | | | | | | |
| Programming no | tes: A by | y-subject listing o | f demographic char | acteristic | s including: | | | | | | |
| | | Treatment | | | | | | | | | |
| | | Subject | | | | | | | | | |
| | | Date of visit | | | | | | | | | |
| | | Date of birth | | | | | | | | | |
| | | Age | | | | | | | | | |
| | | Gender | | | | | | | | | |
| | | Race / Ethnic C | Origin | | | | | | | | |
| | | Height (if collec | cted only once durin | g the stu | dy) | | | | | | |
| | | Weight (if colle | cted only once durin | ig the stu | dy) | | | | | | |
| | | Smoking Histor | y | | | | | | | | |
| | | Alcohol Consur | nption | | | | | | | | |
| | | Xanthine | | | | | | | | | |
| | | Additional stud | y-specific demograp | hy chara | cteristics inclu | ided on the CRF | 7 | | | | |

Sponsor code: DNDI-EMO-03

#### Template L\_CM1\_PG

Listing 16.2.x.xx Listing of Concomitant Medications

| | | ATC Class/ | Drug Name/ | Dose/ | Date/time Started/ | Time Since Last | Started Pre- | Ongoing |
|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Medication Code* | Indication | Freq/Route | Date Stopped | Dose | Trial? | Medication? |

Coded using WHODrug Global version xx.x\*

Programming notes: \* only include this column and the footnote if coding used

Include dose and units (e.g. 5 mg)/Freq/Route

#### Template L\_EX1\_PG

Listing 16.2.x.xx Listing of Exposure Data

| | | | | Dur- | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Start Date/ | Stop Date/ | ation | | Dose | Formulation | / |
| Treatment | Subject | Start Time of Dose | Stop Time of Dose | (days) | Dose | Unit | Route | Frequency |
| Treatment 1 | 1001 | 01JAN2002 | 15FEB2002 | 46 | 25 | mg | Tablet/ | 2xday |
| | | 23:59 | 15:30 | | | | Oral | |

Sponsor code: DNDI-EMO-03

#### Template L\_PK1\_PG

Listing 16.2.4.xx Listing of Emodepside Plasma Pharmacokinetic Concentration-Time Data

| | | {Add. | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | time | | | Planned | Actual time | Time Deviation | Time | |
| Treatment | Subject | var.} | Date | Study Day | Relative Time | (hh:mm) | (min) | (hh:mm) | Concentration (units) |

Below the Limit of Quantification (BLQ) is < xx units (e.g. 1 ng/mL)

Programming notes: Values below LLOQ are shown as BLQ

#### Template L\_PK4\_PG

Listing 16.2.4.xx Listing of Derived Emodepside Pharmacokinetic Parameters

| | | {Add. | | | | | |
|---|---|---|---|---|---|---|---|
| | | time | $AUC_{inf}$ | $AUC_t$ | $C_{max}$ | t <sub>1/2</sub> | $t_{max}$ |
| Treatment | Subject | var.} | (units) | (units) | (units) | (units) | (units) |

Programming notes: Continue with all parameters

Sponsor code: DNDI-EMO-03

#### Template L\_AE1\_PG

Listing 16.2.x.xx Listing of All Adverse Events

| | | | Outcome/ | | | Frequency/ | Related to Study |
|---|---|---|---|---|---|---|---|
| | | System Organ Class / | Onset Date/Time/ | | Severity/ | Action Taken (1)/ | Drug/ |
| | | Preferred Term/ | Resolved Date/Time/ | Time Since Last | Serious/ | Other Action | Treatment |
| Treatment | Subject | Verbatim Text | Duration | Dose | Withdrawal | Taken | Emergent? |
| Treatment 1 | 1001 | Gastrointestinal Disorders / | Resolved/ | 10d 7h 3m | Mild/ | Intermittent/ Dose | Possibly/ |
| | | Intestinal Spasm / | 24SEP2003 13:05/ | | No/ | not changed/ | Yes |
| | | Entero-spasm | 27OCT2003 7:50/ | | Yes | None | |
| | | | 34d 4h 5m | | | | |

<sup>(1)</sup> Action Taken with Study Treatment

Programming notes: For the listing of "other significant AEs" include (from ICH E3) AEs leading to withdrawal, AEs leading to dose reduction (including drug withdrawn, interrupted, reduced or similar) and AEs with AEOSE=Y. If AEOSE has not been collected then use "Otherwise significant" in the CRF.

Sponsor code: DNDI-EMO-03

#### Template L\_LB1\_PG

Listing 16.2.x.xx Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance

| | | | Planned<br>Relative | | Study | | | | | Clinically |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Laboratory test (units) | Time | Date/Time | Day | Value | Reference Interval | RI | BL | Significant? |
| Treatment 1 | 1001 | Alk Phos (U/L) | Time 1 | 01JAN2002 | -1 | 64.00 | 32.0 - 92.0 | | | |
| | | | | 13:34 | | | | | | |
| | | | Time 2 | 01APR2002 | 85 | 84.00 | 32.0 - 92.0 | | | |
| | | | | 07:22 | | | | | | |
| | | ALT (U/L) | Time 1 | 01JAN2002 | -1 | 29.00 | 10.0 - 40.0 | | | |
| | | | | 18:56 | | | | | | |
| | | | Time 2 | 01APR2002 | 85 | 70.00 | 10.0- 40.0 | Н | - 1 | Υ |
| | | | | 09:22 | | | | | | |

RI for Reference Interval flag, BL for Change from Baseline flag;

H = Above reference interval, L = Below reference interval, I = Increase from baseline greater than pre-defined limit, D = Decrease from baseline greater than pre-defined limit

Programming notes: Lists only double-flagged subjects

Sponsor code: DNDI-EMO-03

#### Template L\_LB2\_PG

Listing 16.2.x.xx Listing of All Clinical Chemistry Laboratory Data for Subjects with PCI Abnormalities

| | | Planned<br>Relative | | Alkaline Ph | osphatase (IU, | | Alanine Aı | mino Trans<br>(IU/L) | ferase | Aspartate | Amino Trai | nsferase | Total B | ilirubin (UN | MOL/L) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Time | Date/Time | Result | RI B | L R | esult | RI | BL | Result | RI | BL | Result | RI | BL |
| | | Planned<br>Relative | | Chlorid | le (MMOL/L) | | Gluco | se (MMOL/ | <b>′</b> L) | Potas | sium (MMC | DL/L) | Sodi | um (MMO | ·L/L) |
| Treatment | Subject | Time | Date/Time | Result | RI B | IL R | esult | RI | BL | Result | RI | BL | Result | RI | BL |
| | | | Planned<br>Relative | | Cal | cium (MM | OL/L) | | Creatinin | e (UMOL/L) | | | Etc. | | |
| | Treatm | ent Subject | Time | Date/Time | Result | RI | BL | Resu | lt | RI BL | Resi | ult | RI BL | | |

RI for Reference Interval flag, BL for Change from Baseline flag;

H = Above reference interval, L = Below reference interval, I = Increase from baseline greater than pre-defined limit, D = Decrease from baseline greater than pre-defined limit

Programming notes: Lists only double-flagged subjects

*Include all parameters for the study following the order from the lab report (above is a guide only)* 

Sponsor code: DNDI-EMO-03

#### Template L\_URI\_PG

Listing 16.2.x.xx Listing of Urinalysis Data

| - | Planned | | | Specific Gravity | | рН | | Protein | | Gluco | Glucose |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Relative | | | | | | | | | | | |
| Treatment | Subject | Time | Date/Time | Result | RI | Result | RI | Result | RI | Result | RI |

RI for Reference Interval flag, H = Above reference interval, L = Below reference interval, A = Abnormal result

Programming notes: Include all parameters for the study following the order from the lab report (above is a guide only)

#### Template L\_VS1\_PG

Listing 16.2.x.xx Listing of Vital Signs of Potential Clinical Importance

| | | | | Systolic | Diastolic | |
|---|---|---|---|---|---|---|
| | | Planned Relative | | <b>Blood Pressure</b> | Blood Pressure | Etc |
| Treatment | Subject | Time | Date/Time | (mmHg) | (mmHg) | (units) |
| | | 24 H | 26SEP2012:09:57 | 63 | 148* | |

<sup>\*</sup> Value of potential clinical importance

Sponsor code: DNDI-EMO-03

#### Template L\_EG1\_PG

Listing 16.2.x.xx Listing of ECG Values of Potential Clinical Importance

| | | | | | | | | QT Int. | QT Int. (msec) | | QTcB (msec) | | QTcF (msec) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Heart | | QRS | QRS | | Change | | Change | | Change |
| | | Planned | | Rate | PR Int. | Dur. | Axis | | from | | from | | from |
| Treatment | Subject | Relative Time | Date/Time | (bpm) | (msec) | (msec) | (deg) | Observed | Baseline | Observed | Baseline | Observed | Baseline |
| | | 24 H | 26SEP2012:09:57 | 63 | 148 | 78 | 50 | 390 | 32.7 * | 399 | -27.7 | 396 | -6.5 |

Programming notes: Do not list RR

#### Template L\_EG2\_PG

Listing 16.2.x.xx Listing of Abnormal ECG Findings

| | Pla | | Comment on Clinical | | |
|---|---|---|---|---|---|
| Treatment S | Subject | Time | Date/Time | ECG Finding | Significance |

Programming notes: Lists only values with Normal variant='No' or with comment on ECG result

ECG Finding contains Physician's Opinion from CRF and relates to whole trace (not individual parameters), e.g. Normal, Abnormal - NCS or Abnormal - CS

<sup>\*</sup> Value of potential clinical importance

Sponsor code: DNDI-EMO-03

#### Template L\_PE1\_PG

Listing 16.2.x.xx Listing of Abnormal Physical Examination Findings

Planned Relative

Treatment Subject Time Date/Time Site Details

Programming Notes: List only findings with an 'abnormal' result.

If subjects have multiple abnormal sites at a given time, create a separate row for each site.

#### Template L\_NE1\_PG

Listing 16.2.x.xx Listing of Abnormal Neurological Examination Findings

Planned

Treatment Subject Relative Time Date/Time Type Assessment Details

Programming Notes: Type = (Mental Status, Cranial Nerves, etc.)

List only findings with an 'abnormal' result.

If subjects have multiple abnormal assessment at a given time, create a separate row for each assessment.

# **Appendix A: Laboratory Ranges**

## Pre-determined Changes for Laboratory Data (from FL140 v3)

| | | | | Delta | Delta ranges |
|---|---|---|---|---|---|
| Test | <b>Test Code</b> | Unit | Sex | Acceptable decrease | Acceptable increase |
| Activated partial thromboplastin time | APTTT | sec | Both | - 8.0 | + 8.0 |
| Alanine transferase | ALTN | IU/L | F | - | + 30 |
| Alanine transferase | ALTN | IU/L | M | - | + 30 |
| Albumin | ALB | g/L | Both | - 8 | + 8 |
| Alkaline phosphatase | ALPN | IU/L | Both | - 30 | + 30 |
| Amylase | AMY | U/L | Both | - | + 150 |
| Aspartate transferase | ASTN | IU/L | F | - 30 | + 30 |
| Aspartate transferase | ASTN | IU/L | M | - 30 | + 30 |
| Basophils | BASO | 10 <sup>9</sup> /L | Both | - | + 0.30 |
| Bilirubin conjugated | DBIL | μmol/L | Both | - | + 4.0 |
| Bilirubin total | TBIL | μmol/L | F | - 20.0 | + 10.0 |
| Bilirubin total | TBIL | μmol/L | M | - 20.0 | + 10.0 |
| Bilirubin unconjugated | IBIL | μmol/L | Both | - | - |
| C-reactive protein | CRP | mg/L | Both | - | - |
| CK relative index | CKMBR | % | Both | - | - |
| Calcium | CA | mmol/L | Both | - 0.4 | + 0.4 |
| Carbon dioxide | CO2 | mmol/L | Both | - 8 | + 8 |
| Chloride | CL | mmol/L | Both | - 10 | + 10 |
| Cholesterol | CHOL | mmol/L | Both | - | + 0.7 |
| Creatine kinase | CK | IU/L | F | - | + 400 |
| Creatine kinase | CK | IU/L | M | - | + 400 |
| Creatinine | CREA | μmol/L | Both | - | + 40 |
| Creatinine (DOA urine) | CREDA-U | mmol/L | Both | - | - |
| Eosinophils | EOS | 10 <sup>9</sup> /L | Both | - | + 0.50 |
| Erythrocyte sedimentation rate | ESR | mm/h | Both | - | = |
| Fibrinogen | FIB-C | g/L | Both | - | - |
| Free T3 | FT3 | pmol/L | Both | - 3.5 | + 3.5 |
| Free T4 | FT4 | pmol/L | Both | - 15.0 | + 15.0 |
| Gamma glutamyl transferase | GGT | IU/L | F | - | + 40 |
| Gamma glutamyl transferase | GGT | IU/L | M | - | + 40 |
| Globulin | GLOB | g/L | Both | - 8 | - |
| Glucose | GLU | mmol/L | Both | - 1.5 | + 2.5 |
| Haematocrit | НСТ | L/L | Both | - 0.050 | - |
| Haemoglobin | НВ | g/L | Both | - 20 | - |
| High density lipoprotein | HDL | mmol/L | Both | - 1.50 | + 1.50 |
| International normalised ratio | INRR | ratio | Both | - | - |
| Lactate dehydrogenase | LDH | IU/L | Both | - | + 150 |
| Lymphocytes | LYMP | 10 <sup>9</sup> /L | Both | - 1.50 | + 1.50 |
| Magnesium | | 1 | ъ л | 1 | |
| | MG | mmol/L | Both | - | - |
| Mean cell haemoglobin | MG<br>MCH | mmol/L pg | Both | - 2.0 | + 2.0 |
| Mean cell haemoglobin Mean cell haemoglobin concentration | | | _ | -<br>- 2.0<br>- 25 | + 2.0<br>+ 25 |

| | | | | Delta ranges | |
|---|---|---|---|---|---|
| Test | Test Code | Unit | Sex | Acceptable decrease | Acceptable increase |
| Monocytes | MONO | 10 <sup>9</sup> /L | Both | - 0.50 | + 0.50 |
| Neutrophils | NEUT | 10 <sup>9</sup> /L | Both | - 2.00 | + 8.00 |
| Phosphate | PHOS | mmol/L | Both | - 1.00 | + 1.00 |
| Platelets | PLT | 10 <sup>9</sup> /L | Both | - 100 | + 100 |
| Platelets (citrate tube) | PLTC | 10 <sup>9</sup> /L | Both | - 100 | + 100 |
| Potassium | K | mmol/L | Both | - 0.8 | + 0.8 |
| Prolactin | PROL | μg/L | Both | - | - |
| Prothrombin time | PTT | sec | Both | - 4.0 | + 4.0 |
| Red blood cells | RBC | 10 <sup>12</sup> /L | Both | - 1.0 | - |
| Reticulocyte | RET | % | Both | - | - |
| Reticulocyte count | RETC | 10 <sup>9</sup> /L | Both | - | - |
| Reticulocyte manual count | RETM | 10 <sup>9</sup> /L | Both | - | - |
| Sodium | NA | mmol/L | Both | - 8 | + 8 |
| Thrombin time | TT | sec | Both | - | - |
| Thyroid stimulating hormone | TSH | mIU/L | Both | - 3.00 | + 3.00 |
| Total protein | TP | g/L | Both | - 15 | - |
| Triglycerides | TG | mmol/L | Both | - | + 1.5 |
| Urea | UREA | mmol/L | Both | - 5.0 | + 2.0 |
| Uric acid | UA | μmol/L | Both | - 100 | + 100 |
| Urine pH | UPH | N/A | Both | - 4 | + 4 |
| Urine red blood cells | URBC | 10 <sup>6</sup> /L | Both | - | + 10 |
| Urine white blood cells | UWBC | $10^{6}/L$ | Both | - | + 100 |
| White blood cells | WBC | 10 <sup>9</sup> /L | Both | - 2.0 | + 8.0 |

## **Appendix B: Pharmacokinetic Analysis**

### 1 Calculation Methods

## 1.1 Data Handling Conventions

#### 1.1.1 Actual vs Planned Times

Actual sample times will be used for the calculation of pharmacokinetic parameters and for individual concentration-time plots.

Planned sampling times will be used to calculate the concentration-time summary statistics and summary concentration-time plots.

#### 1.1.2 Missing and BQL Concentrations

Missing values will not be used in any way.

For calculation of all pharmacokinetic parameters and individual profile plots, plasma concentrations below the quantifiable limit (BQL) of the assay will not be used for the calculation of PK parameters (except BQL values observed at time points before the maximum concentration, which will be taken as zero).

BQL values observed post dose will be substituted by one half of the lower limit of quantification for calculation of plasma concentration summary statistics. Pre dose values will be taken as zero. The number of imputed values will be included in the summary table.

## 1.2 AUC Calculations

The AUC will be calculated by a combination of linear and logarithmic methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations

#### 1.3 Lambda-z Calculations

The apparent terminal phase rate-constant ( $\lambda_z$ ) will be estimated by linear regression of logarithmically transformed concentration versus time data. Only those data points

which are judged to describe the terminal log-linear decline will be used in the regression.

During the analysis, repeated regressions are carried out using the last three points with non-zero concentrations, then the last four points, last five, etc. Points prior to  $C_{max}$  are not used. Points with a value of zero for the concentration are excluded. For each regression, an adjusted  $R^2$  is computed. The  $\lambda_z$  using the regression with the largest adjusted  $R^2$  is selected. If the adjusted  $R^2$  does not improve, but is within 0.0001 of the largest adjusted  $R^2$  value, the regression with the larger number of points is used.  $\lambda_z$  must be positive, and calculated from at least three data points.

For non-compartmental analysis uniform weighting will be applied.

#### 1.4 Observed v Predicted Values

For parameters dependent on  $\lambda_z$ , the 'predicted' rather than the 'observed' parameters will be calculated.

The 'predicted' parameters are calculated using  $\hat{C}_t$  (the predicted value of the concentration at time tn); whilst the 'observed' parameters use the last observed concentration.

## 2 General Considerations for Data Analysis

#### 2.1 Derived and transformed data

In general, concentration and concentration-related quantities, rate constants and half-lives (e.g.  $C_{max}$ , AUC,  $t_{1/2}$  and MRT) will be analysed after logarithmic transformation. Logarithmic transformations will use natural logarithms (log<sub>e</sub>). A list of those parameters that will be log transformed are given below.

## 2.2 Summary data

Means at any time will only be calculated if at least 2/3 of the individual data are measured and are above the lower of quantification (LLOQ).

# 3 Parameter Definitions

## 3.1 Plasma Parameters

## 3.1.1 Emodepside

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| Concentrations and | times | | | • | | - Cu | · |
| C <sub>max</sub> | Maximum (peak) plasma concentration | The maximum (peak) plasma concentration will be obtained directly from the concentration-time data. | ng/mL | Y | Cmax | CMAX | $C_{max}$ |
| C <sub>max</sub> /Dose | Dose-normalised C <sub>max</sub> to infinity | The dose-normalised $C_{max}$ will be calculated as $C_{max}$ /Dose administered | (ng/mL)/mg | Y | Cmax_D | CMAXD | C <sub>max</sub> /D |
| C <sub>max,norm</sub> | Observed maximum plasma concentration corrected by dose and body weight | The C <sub>max</sub> normalised by dose and body weight will be calculated as C <sub>max</sub> /(Dose administered*body weight) | (ng/mL)/(mg*kg) | Y | N/A | CMAXWD | $C_{\text{max,norm}}$ |
| t <sub>max</sub> | Time to reach maximum (peak) plasma concentration | The first time of maximum (peak) plasma concentration will be obtained directly from the concentration-time data. | h | N | Tmax | TMAX | t <sub>max</sub> |
| Half-life | | | | | | | |
| $\lambda_z$ | Terminal rate constant | The apparent terminal phase rate-constant $(\lambda_z)$ will be estimated by linear regression of logarithmically transformed concentration versus time data. | 1/h | Y | Lambda_z | LAMZ | $\lambda_{\mathrm{z}}$ |
| Point terminal | Number of points for<br>Lambda z | The number of time points used in calculating Lambda z | - | - | No_points_lambda<br>z | LAMZNPT | $n_{pts}$ |
| t <sub>½,0-7d</sub> | Terminal half-life | The terminal half-life calculated from the terminal slope of the log concentration-time curve, as follows: $t_{1/2} = \frac{\log_e 2}{\lambda_z}$ | h | Y | HL_Lambda_z | LAMZHL | t <sub>1/2,0-7d</sub> |
| t½,0-24h | Dominant half-life | The half-life calculated from the terminal slope of the log concentration-time (0-24h) curve, as follows: $t_{1/2} = \frac{\log_e 2}{\lambda_z}$ | h | Y | HL_Lambda_z | LAMZHLD | t <sub>1/2,0-24</sub> |

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| Areas under the cur | | | 1 | | | 1 | |
| AUC <sub>last</sub> | Area under the plasma<br>concentration-time curve<br>from time zero to time of last<br>measurable concentration | The area under the concentration-time curve from zero time (pre-dose) to the time of last quantifiable concentration will be calculated using the (specified) trapezoidal method. | h*ng/mL | Y | AUC_last | AUCLST | AUC <sub>last</sub> |
| AUC <sub>0-7d</sub> | Area under the plasma concentration-time curve from time zero to 7 days | The area under the concentration-time curve from zero time (pre-dose) to 7 days will be calculated using the (specified) trapezoidal method. If $\lambda_z$ is not estimable, a partial AUC is not calculated (when $t_{last} < t$ ). | h*ng/mL | Y | User specified area | AUCINT | $\mathrm{AUC}_{7\mathrm{d}}$ |
| AUC <sub>0-7d</sub> /Dose | Dose-normalised AUC from time zero to 7 days | The dose-normalised AUC from time zero to 7 days will be calculated as AUC <sub>0-7d</sub> /Dose administered | (h*ng/mL)/mg | Y | N/A | AUCINTD | AUC <sub>7d</sub> /D |
| AUC <sub>0-7d,norm</sub> | Area under the concentration-time curve from time zero to 7 days corrected by dose and body weight | The AUC from time zero to 7 days normalised by dose and body weight will be calculated as AUC <sub>0-7d</sub> /(Dose administered*body weight) | (h*ng/mL)/(mg*kg) | Y | N/A | AUCINTWD | AUC7d,norm |
| Clearance, volume | of distribution and mean residen | ce time | | | | | |
| MRT <sub>last</sub> | Mean Residence Time | The mean residence time will be calculated using: $MRT = \frac{AUMC_{last}}{AUC_{last}}$ | h | Y | MRTlast | MRTEVLST | $MRT_{last}$ |

Sponsor code: DNDI-EMO-03

# **Appendix C: Sample Page Layout**

| DNDi: DNDI-EMO-03 Part 1 | | |
|---|---|---|
| Population: [Pop] | | |
| | | · |
| | Table [number] [title] | |
| | Column headers | _ |
| | Main body of output | _ |
| | Source: Listing [16.2.xx] | _ |
| Footnotes about the table or list | ing text go here. | |
| Program: [Prog Name] | [Date] | <br>HMR 17-008 Part 1 |
| Produced By:[Username] | | |

\*y = last page of individual output Font size will be Arial 9.5pt. The following margins will be used: Left: 1", Right: 1", Top: 1", Bottom: 1"